CLINICAL TRIAL: NCT07406698
Title: Strategic Timing of Endoscopic Procedural Interventions in Infected Necrotizing Pancreatitis: The STEP-IN Trial
Brief Title: Strategic Timing of Endoscopic Interventions in Infected Necrotizing Pancreatitis
Acronym: STEP-IN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2401309
Record Dates: First submitted 2026-02-02; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Pancreatitis, Acute Necrotizing
Keywords: Endoscopic ultrasound; Drainage; Necrotic collection; Timing of intervention
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early endoscopic intervention in infected necrotizing pancreatitis (Active Comparator): In the early treatment group, EUS-guided drainage is undertaken within 72 hours of randomization, earlier than 28 days after the onset of acute pancreatitis.
  Interventions: Procedure: EUS-guided transluminal drainage of necrotic collection
- Postponed endoscopic intervention in infected necrotizing pancreatitis (Active Comparator): In the postponed treatment group, EUS-guided drainage is undertaken only from 28 days after the onset of acute pancreatitis when the collection is fully or predominantly walled-off (encapsulated).
  Interventions: Procedure: EUS-guided transluminal drainage of necrotic collection

INTERVENTIONS:
Procedure: EUS-guided transluminal drainage of necrotic collection — EUS-guided drainage of the necrotic collection is performed by placement of a metal stent within the dominant collection.

SUMMARY:
Pancreatic necrosis complicates approximately 20-30% of severe acute pancreatitis cases. While many collections resolve without intervention, persistent symptomatic collections-particularly when infected-are associated with significant morbidity and mortality and frequently require procedural management. Current guidelines recommend delaying intervention until collections are fully walled off, typically around four weeks. However, in clinical practice, many patients deteriorate before this window is reached.

Prospective data from our institution, supported by recent meta-analyses, suggest that early intervention using modern endoscopic techniques can be performed safely, even when undertaken within the first four weeks of disease onset. We believe that, in appropriately selected patients, early endoscopic intervention may prevent clinical deterioration, reduce complications, shorten hospital stay, and decrease overall healthcare utilization compared with a delayed approach.

To formally evaluate this strategy, an international, multicenter randomized trial is being conducted, entitled Strategic Timing of Endoscopic Procedural Interventions in Infected Necrotizing Pancreatitis (STEP-IN Trial).

DETAILED DESCRIPTION:
Acute pancreatitis imposes a significant burden on the US health-care system, resulting in approximately 300,000 hospital admissions annually and generating costs exceeding $2 billion. Necrotizing pancreatitis develops in approximately 20 to 30% of patients with acute pancreatitis. It can mature into a contained necrotic collection, typically four weeks into the disease course. While some collections may resolve without an intervention, persistent collections can result in symptoms such as pain, abdominal fullness restricting nutrition, vomiting due to gastric outlet obstruction, obstructive jaundice due to a large collection in the pancreatic head, new-onset or persisting organ failure, continued unwellness or infection that is associated with a mortality of 15-20%, and requires drainage and necrosectomy.

International guidelines recommend that, when possible, treatment should be delayed in patients with suspected or confirmed infected necrotizing pancreatitis, to allow for the collection to be walled-off with better demarcation and liquefaction of the necrosis, which generally takes around 4 weeks. The main rationale for postponement of an invasive intervention is to prevent complications, but this rationale originated from an era when open surgical necrosectomy was performed.

Recently, there has been a shift away from open surgery towards minimally invasive treatment approaches. The current standard approach for treatment is a minimally invasive step-up approach with percutaneous catheter or transluminal endoscopic drainage as the first step, followed by video-assisted retroperitoneal/sinus-tract or transgastric necrosectomy. The development of cautery-enhanced lumen-apposing metal stents (LAMS) for endoscopic drainage has significantly simplified the technical aspects of the procedure that facilitates its performance even in very sick patients.

Although international guidelines recommend postponing treatment until 4-weeks when the necrosis is better demarcated, in an international survey of expert pancreatologists, 45% of the respondents reported that they recommend immediate catheter drainage as soon as infected pancreatic and peripancreatic necrosis is diagnosed. In addition, a recent clinical practice guideline from the American Gastroenterological Association states that catheter drainage should be strongly considered when there is a concern of infection, even in the early phase of disease. However, a multicenter, randomized trial did not show superiority for immediate over postponed catheter drainage in reducing complications in patients with infected necrotizing pancreatitis.

Prospective data from our institution and from the meta-analysis suggest that interventions can be undertaken safely adopting state-of-the-art endoscopic methods even when the onset of pancreatitis is less than 4 weeks. Our data also suggest that although a significant proportion of patients undergoing early interventions (adopting an endoscopic approach) do not have a fully encapsulated collection, their treatment outcomes are not negatively impacted by such approach. If an early intervention, adopting an endoscopic approach, can be undertaken safely, it potentially can prevent further clinical deterioration and therefore complications, decrease length of hospitalization as patients may not have to wait for 3 to 4 weeks and overall treatment costs as compared to postponing the intervention until 4-weeks when the necrosis is fully walled-off.

The STEP-IN trial therefore is a natural step in the advancement of our understanding of timing of interventions in necrotizing pancreatitis as it answers an important clinical question: can early interventions be undertaken safely without subjecting patients to an arbitrary time frame of 4-weeks? In this study we challenge the existing paradigm of delayed intervention in attempt to further improve the clinical outcomes in patients with infected necrotizing pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with symptomatic necrotic collection diagnosed on MRI or CT abdomen/pelvis, defined as fluid collection in the setting of documented pancreatic necrosis that contains necrotic material and encased within a partial or complete wall.
3. Documented or suspected infected necrotizing pancreatitis 1) Documented infected necrotizing pancreatitis, defined as: i. Positive culture obtained with percutaneous fine needle aspiration from the pancreatic necrotic collection (if intervention is undertaken ≤14 days of onset of acute pancreatitis) ii. OR gas in the necrotic collection on imaging at any time. 2) Suspected infected necrotizing pancreatitis, if >14 days after onset of disease, defined as: i. Persistent organ failure in patients admitted to the ICU ii. OR presence of at least three of the following six clinical/laboratory parameters (SIRS criteria or elevated CRP or elevated procalcitonin) with no other infection focus. These clinical criteria are considered sufficiently reliable only after the initial 14 days of acute pancreatitis:

   1. Temperature >100.4 °F or <96.8 °F
   2. Heart rate > 90 beats/min
   3. Respiratory rate >20 breaths/min or PaCO2 < 32 mmHg
   4. WBC count >12,000/mm³, or <4,000/mm³, or more than 10% immature band cells
   5. CRP ≥ 30mg/L
   6. Procalcitonin ≥ 1ng/mL
4. Endoscopic drainage of the necrotic collection is technically feasible as deemed by the treating physician.

Exclusion Criteria:

1. Age < 18 years
2. > 26 days after the onset of acute pancreatitis
3. Indication for emergency laparotomy for abdominal catastrophe (e.g. bleeding, bowel perforation, abdominal compartment syndrome).
4. Necrotic collection is not amenable for endoscopic intervention.
5. Pregnancy.
6. Unable to obtain informed consent from the patient or legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of major complications or death | 6 months
  Proportion of patients experiencing a major complication or death. Major complications comprise new onset organ failure, new onset systemic dysfunction, enteral or pancreatic-cutaneous fistula, intraabdominal bleeding, or visceral perforation.

SECONDARY OUTCOMES:
Mortality | 6 months
  Proportion of patients with mortality from any cause
Major complications | 6 months
  Proportion of patients experiencing major complications. Major complications comprise new onset organ failure (respiratory, cardiovascular, renal, gastrointestinal, hepatic, hematologic, neurologic, or metabolic failure), new onset systemic dysfunction, enteral or pancreatic-cutaneous fistula, intraabdominal bleeding, or visceral perforation
New onset single and multiple organ failure | 6 months
  Proportion of patients with new onset failure of at least one organ system
New onset systemic dysfunction | 6 months
  Proportion of patients with worsening of any pre-existing medical condition
Enterocutaneous and pancreatic fistula | 6 months
  Proportion of patients with enterocutaneous fistula or pancreatic fistula. Enterocutaneous fistula is the formation of a fistula between the small bowel or colon and skin as indicated by feculent output from a percutaneous catheter or surgical wound site, confirmed on imaging or surgery.
  Pancreatic fistula is the formation of a fistula between the pancreas and skin as indicated by amylase-rich fluid output from a percutaneous catheter or surgical wound site, persisting after 3 months, and requiring specific treatment that include parenteral or enteral nutrition, antibiotics, somatostatin analogues and minimally invasive drainage.
Intraabdominal bleeding | 6 monthts
  Proportion of patients with intraabdominal bleeding. Intraabdominal bleeding is defined as bleeding within the intraabdominal cavity or gastrointestinal tract requiring interventional procedure
Visceral perforation | 6 months
  Proportion of patients with visceral perforation. Visceral perforation is defined as the perforation of a visceral organ requiring interventional procedure
Incisional hernia | 6 months
  Proportion of patients with incisional hernia. Incisional hernia is defined as herniation of intraabdominal structures through an area of weakness in the abdominal fascia, requiring surgical intervention or persisting at 6-month follow-up
Surgical site infection | 6 months
  Proportion of patients with surgical site infection. Surgical site infection is defined as the infection in superficial or deep layers of the abdominal wall at the site of prior intervention, as evident by the presence of purulent drainage or abscess on physical examination, imaging and/or requiring intervention
New onset diabetes | 6 months
  Proportion of patients with new onset diabetes. New onset diabetes is defined as new onset elevation in fasting plasma glucose ≥ 126 mg/dL, 2-hour plasma glucose ≥ 200 mg/dL after an oral glucose tolerance test or HbA1c ≥ 6.5%
New diagnosis of exocrine pancreatic insufficiency | 6 months
  Proportion of patients with new diagnosis of exocrine pancreatic insufficiency. Exocrine pancreatic insufficiency is defined as fecal elastase level < 200μg/g in patients not previously taking pancreatic enzyme supplements
Procedure-related adverse events | 6 months
  Proportion of patients with any adverse event resulting from endoscopic or surgical intervention
Disease-related adverse events | 6 months
  Proportion of patients with any adverse event resulting from necrotizing pancreatitis
Number of interventions | 6 months
  Number of interventions performed for treatment of infected necrotizing pancreatitis including endoscopic, surgical and radiological interventions
Length of hospitalization | 6 months
  Length of hospitalization, including length of ICU stay
Readmissions | 6 months
  Proportion of patients with hospital admissions due to underlying disease or procedure-related adverse events
Presence of systemic inflammatory response syndrome (SIRS) at 72 hours post-index intervention | 72 hours
  Proportion of patients with positive SIRS at 72 hours post-index procedure. Positive SIRS is defined by the presence of at least two of the following four criteria:
  1. Body temperature >100.4 °F or < 96.8 °F
  2. Heart rate > 90 beats/minute
  3. Respiratory rate > 20 breaths/minute or PaCO2 < 32mmHg
  4. White blood cell count > 12 or < 4 x109/L or > 10% immature neutrophils
New onset systemic inflammatory response syndrome (SIRS) at 72 hours post-index intervention | 72 hours
  Proportion of patients with new onset SIRS at 72 hours post-index intervention. Positive SIRS is defined by the presence of at least two of the following four criteria:
  1. Body temperature >100.4 °F or < 96.8 °F
  2. Heart rate > 90 beats/minute
  3. Respiratory rate > 20 breaths/minute or PaCO2 < 32mmHg
  4. White blood cell count > 12 or < 4 x109/L or > 10% immature neutrophils
Resolution and improvement of systemic inflammatory response syndrome (SIRS) at 72 hours post-index intervention | 72 hours
  Proportion of patients with resolution of SIRS at 72 hours post-index intervention. Positive SIRS is defined by the presence of at least two of the following four criteria:
  1. Body temperature >100.4 °F or < 96.8 °F
  2. Heart rate > 90 beats/minute
  3. Respiratory rate > 20 breaths/minute or PaCO2 < 32mmHg
  4. White blood cell count > 12 or < 4 x109/L or > 10% immature neutrophils
Technical success | 6 months
  Rate of technical success. Technical success is defined as the successful completion of EUS-guided drainage of the necrotic collection
Treatment success | 6 months
  Rate of treatment success. Treatment success is defined as the resolution of necrotic collection on CT scan in association with clinical resolution of symptoms at 6 months from index intervention
Health-related quality of life (HRQoL) | 6 months
  Health-related quality of life (HRQoL) scores as assessed by the Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36)
Overall treatment costs | 6 months
  Overall treatment costs from admission until hospital discharge. All relevant costs pertaining to treatment will be taken into consideration - procedure costs, cost of inpatient hospital stay (from date of procedure to discharge), cost of medications, cost of materials, cost of anesthesia, cost of pharmacy and cost of imaging studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health Digestive Health Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No